CLINICAL TRIAL: NCT02405806
Title: Clinical Effects of Nutrition on Metabolic Risk Factors and Mechanisms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Bodil Ohlsson, Professor, senior consultant, Region Skane
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 140917-281
Record Dates: First submitted 2015-02-23; First posted 2015-04-01 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Obesity; Diet Modification
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- low carbohydrate food (Experimental): The subjects will be given a diet with moderate, low carbohydrate content for 3 months, or as a single test meal, and this will be evaluated in metabolic parameters, microbiota and biomarkers in serum as described previously.
  Intervention: Food: Low carbohydrate food
  Interventions: Dietary Supplement: low carbohydrate food
- standard food (Active Comparator): The subjects will be given a diet with standard food as a single test meal, and this will be evaluated in metabolic parameters, microbiota and biomarkers in serum, as described Intervention: Food: Standard food
  Interventions: Dietary Supplement: standard food

INTERVENTIONS:
Dietary Supplement: low carbohydrate food — low carbohydrate food
  Arms: low carbohydrate food
Dietary Supplement: standard food — standard food
  Arms: standard food

SUMMARY:
The overall aim for this study is to evaluate the clinical effects of a modified diet on metabolic risk factors such as diabetes mellitus and obesity, and the mechanisms this nutrition composition exerts on gastrointestinal physiology, inflammatory responses, and quality of life, where the subjects are their own controls.

Within this study, the investigators will be able to relate the nutritional composition to metabolic disorders, the gut microbiota, secreted intestinal neuropeptides, and bio- and inflammatory markers in serum, plasma and urine.

DETAILED DESCRIPTION:
Material and Methods

Subjects are recruited consequently from the primary care, and from the Department of Endocrinology.

Study population

The investigator will include:

1. patients with type 2 diabetes to study the effect of a modified diet for 3 months;
2. healthy volunteers for intake of two different breakfasts with some days in between the meals.

All categories will be exposed to exactly the same study design.

Protocols:

Various protocols will be used in the study, to collect information about the status at inclusion, and to be able to measure changes in anthropometry, health status and symptoms during the study period.

Study-questionnaire:

This questionnaire is similar to the questionnaires used in the great population cohorts Malmö Diet and Cancer Study (MDCS, general population from Malmö, N = 28 000), and Malmö Offspring Study (MOS) (general population from Malmö, children and grandchildren to participants in MDCS, calculated to include 5000 participants, started 2013, supported by grants from VR). It is also used in a newly started endoscopy study where all consecutive patients performing a colonoscopy at the Department of Gastroenterology in Malmö will be included (calculated to include 2000 participants). The questionnaire contains questions about socioeconomic factors, life style factors (including diet, smoking, stuff use, alcohol habits, physical activity), medical health, drug consumption, heredity factors and gastrointestinal symptoms.

Nutrition questionnaire:

This questionnaire is used to get information about ordinary diet, energy intake, and so on. This basic information is used to plan the diet from Life Science Lab, so similar energy supply and breakfast are provided.

36-item Short-Form questionnaire (SF-36): This is a world-wide used instrument to evaluate quality of life. It has been used to measure quality of life in many various diseases, and norm value references are available. The instrument measures physical functioning, role functional-physical, bodily pain, general health, vitality, social functioning, role functioning-emotional, and mental health. These parameters are valuable to evaluate, to estimate the effects evoked in daily life, by a change in life style factors.

Anthropometric protocol:

This questionnaire is used to screen the study participants before inclusion, and to be able to exclude patients with already ongoing weight-reducing diet. In addition, it contains questions about BMI, body composition, and a basal physical examination.

Satiety scoring:

This protocol has been used in previous studies by the group, to estimate the degree of hunger/satiety before and after a standardized meal.

Nutrition:

All subjects will get the diet delivered free from charge from Life Science Lab (Lund University). Life Science Lab was founded 1998 as a leading medical and technical research for advanced cardiovascular and thoracic surgery sciences. Due to the importance of life style effects on the cardiovascular diseases and well-being, Life Science Lab also conducts life style-related science to reduce known risk factors for cardiovascular diseases. The main focus is to develop healthy nutrition in normal food formula by reforming the food-meal composition for everyone. The meal-diet consists of ordinary raws, but with minimal industrial processing. The food is based on traditional Nordic raws, e.g. whole grains, vegetables, leguminous, root crops, fat fish, birds, fruits, berries and nuts. At the same time, the amount of sugar, read meat, processed meat, and dairy products is limited. The diet has a good nutritional supply, but contains less calories than what is usually recommended (2000 kcal/day compared with 2400 kcal/day).

The meal is planned together with the kitchen of Life science Lab. Food composition, recipes, and instructions how to cook the food is delivered regularly from Life Science Lab for lunch and dinner. The breakfasts for the subjects are planned together with the PI and the nutritionist at Life Science Lab, but the subjects have to buy the food themselves. Three alternatives are suggested, depending on their ordinary breakfast ingested, described in the nutrition questionnaire.

Neuropeptides/inflammatory markers:

The neuropeptides, or their precursors, that will be studied in serum/plasma are peptides involved in regulation of satiety and digestion, e.g. cholecystokinin (CCK), gastrin, ghrelin, glucagon-like peptide-1 (GLP-1), and glucagon-like peptide-2 (GLP-2), leptin, motilin, neurotensin, oxytocin, and peptide YY (PYY). To evaluate permeability defects in the intestinal mucosa, levels of zonulin and bacterial endotoxins, i.e. lipopolysaccharides, will be measured in plasma. Low-graded inflammation is reflected by high-sensitive C-reactive protein (CRP), plasminogen activator inhibitor type 1 (PAI-1), and factors involved in AGE will be analyzed. In addition, different cytokines, tracers, and routine analyses will be performed. Cooperation with laboratories in Denmark and Great Britain will be established.

Gut microbiota:

DNA extractions and Terminal Restriction Fragment Length Polymorphism (T-RFLP) and quantification of specific bacterial groups will be done by quantitative polymerase chain reaction (PCR) in accordance with the protocols the investigator has used and described earlier by the research group. As reference, a restricted number of samples will be analyzed with massively-parallel pyrosequencing of partial ribosomal ribonucleic acid (rRNA) ribosomal genes. The gut microbiota bacterial constitution (bacterial species) will be correlated to gastrointestinal symptoms and diseases, and changes in bio- and inflammatory markers.

Study Design

When a group of patients are recruited, the investigator will have an information meeting for the whole group. At that meeting, held by the PI, the subjects will receive medical information about metabolic diseases, and about nutrition and its effects on health and disease.

After this initial meeting, the subjects are handled individually. For overview, se flow-chart, last page. At inclusion, all subjects have to complete questionnaires and some examinations:

1. Study-questionnaire containing questions about ordinary lifestyle factors, socioeconomic factors, health- and drug information, heredity, and gastrointestinal symptoms;
2. Nutrition questionnaire containing information about ordinary food habits
3. Quality of life questionnaire SF-36;
4. Anthropometric protocol, including nutritional screening, completed by the investigator; and
5. Eight tubes (SST- phenolsulfotransferase platelet survival time (PST)- and ethylenediaminetetraacetic acid (EDTA) tubes), à 6 ml, to collect serum, plasma and blood cells. Feces sampling for microbiota analyses. Urine sampling during the night. All biological material will be stored at -20 ◦C or -80◦ C for later analyses, or analyzed at once (Hb, leukocytes, thrombocytes, CRP, electrolytes, liver enzymes, lipids, bleeding status, glomerular filtration rate (GFR), insulin, fp-glucose, HbA1c and thyroid-stimulating hormone (TSH), cobalamin, folate and routine urine analyses incl microalbuminuria).

The questionnaires 1, 3, 4, and 5, and experimental procedures will be repeated after 3 months of the diet and at termination after 6 months, with standard food the last 3 months.

Two weeks after introduction of the new diet, insulin, glucose and proinsulin are measured in plasma/serum, along with anthropometric protocol.

During the evaluation of the diet, the subjects have to continue with the same degree of physical activity as previously. No dietary supplements such as fish oil, probiotics or multivitamin drugs are allowed to take. As most one visit to a restaurant or to another diet per week is allowed. Journeys or a stay during a longer time period at another place must be discussed with the leader of the research. Maximal intake of alcoholic beverages is 30 g ethanol/week. 12 g ethanol corresponds to the following: 1 bottle (50cl) ordinary beer, 1 bottle (33cl) strong beer, 1 glass (15cl) wine, 1 glass (8cl) strong wine, or 1 glass (4cl) spirits. formula: volume% x ml volume/100 x 0.8.

Test meal in a substudy of healthy volunteers

The subjects come fasting (12 h) in the morning, bringing the breakfast to consume. Before starting the meal, two blood samples are taken with 10 min in between. After the start of the meal, a new blood sample is collected at 10, 20, 30, 45, 60, 90, 120, and 180 min afterwards. Each blood sample consists of 6 ml plasma. At the same time intervals, the satiety score is completed. With a few days in between, the same procedure is performed where their previous ordinary, daily breakfast is replaced by the new diet, so that 2 test meals are performed during run-in; one with ordinary breakfast and one with new diet breakfast.

During the whole study, PI has a close contact (email and phone) with the patient to be able to support the patient and enhance compliance as much as possible.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects should be healthy.
* Prediabetes should have fasting plasma glucose levels o 5.6-6.9 mmol/l or plasma glucose level 2 h after an oral glucose test of 7.8-11.1 mmol/l, without any diabetes treatment.
* Patients with diabetes should have type-2 diabetes.
* Obesity should have BMI 30-3 and glucose levels within reference values

Exclusion Criteria:

* Patients with diabetes or obesity should not have severe cardiac, kidney, liver or psychiatric diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-11; Primary Completion 2015-10-15 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in metabolic effects, intestinal permeability and microbiota composition after food intervention | 3 months
  In the larger study, the investigator will give the patients a moderate, low carbohydrate food for 3 months and then evaluate the effects in plasma concentration of insulin, fp-glucose, C-peptide, proinsulin, HbA1c, lipids, and zonulin. Feces wil be analyzed for microbiota composition as quantified by PCR.

SECONDARY OUTCOMES:
Quality of life as assessed by the SF-36 | 3 months
  In the larger study, the investigator will give the patients a moderate, low carbohydrate food for 3 months and assess the quality of life before and after intervention by SF-36

OTHER OUTCOMES:
Change from baseline in hormonal effects of food intervention | 3 hours
  The investigator will test one single meal of each food type, standard food or a moderate, low carbohydrate food and then evaluate the plasma concentration over 3 hours of cholecystokinin (CCK), gastrin, ghrelin, glucagon-like peptide-1 (GLP-1), glucagon-like peptide-2 (GLP-2), leptin, motilin, neurotensin, oxytocin, and peptide YY (PYY).

CONTACTS AND LOCATIONS:
Overall Officials: Bodil Ohlsson, Professor, Principal Investigator — Lund University

REFERENCES:
- [Background] Ohlsson B, Bjorgell O, Ekberg O, Darwiche G. The oxytocin/vasopressin receptor antagonist atosiban delays the gastric emptying of a semisolid meal compared to saline in human. BMC Gastroenterol. 2006 Mar 16;6:11. doi: 10.1186/1471-230X-6-11. PMID 16542457
- [Background] Sullivan M, Karlsson J, Taft C. SF-36: Swedish manual and interpretation guide, 2nd Edition. Gothenburg: Sahlgrenska University Hospital. 2002.